CLINICAL TRIAL: NCT06579651
Title: Nailfold Capillaroscopic Pattern Changes and Its Correlation with Interstitial Lung Disease (ILD) in Systemic Sclerosis (SSc) Patients.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennatullah Salaheldin, Mennatullah Salaheldin Mohamed, Assiut University
Other Study IDs: NVC in SSc patients
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Systemic Sclerosis (SSc)
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Microscopic Angioscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Nailfold videocapillaroscopy (NVC) — Nailfold videocapillaroscopy (NVC) is the validated technique to assess SSc microvascular damage and is useful for the early diagnosis and follow-up of SSc micro- angiopathy.

SUMMARY:
Detection of different pattern of nail fold capillary changes in SSc patients. Correlation of nail fold capillary changes in SSc patients with ILD.

DETAILED DESCRIPTION:
SSc is a connective tissue disease characterized by early microvascular damage and dysfunction and immune system activation, as well as progressive fibrosis in the skin and internal organs.

Nailfold videocapillaroscopy (NVC) is the validated technique to assess SSc microvascular damage and is useful for the early diagnosis and follow-up of SSc micro- angiopathy.

Several studies have demonstrated correlations between microvascular damage extent and the severity of internal organ involvement, showing that NVC abnormalities correlate with disease activity and severity and may be also predictive for disease worsening. Furthermore, successful treatments have been shown to reduce NVC abnormalities in SSc cases, and these findings support the importance of NVC in monitoring SSc patients and also suggest its possible role as an outcome measure for microangiopathy in clinical trials.

Three different NVC patterns of microvascular damage have been described ("early" , "active" , "late" ).

ELIGIBILITY:
Inclusion Criteria:

* Adult SSc Patients

Exclusion Criteria:

- 1-SSc patients aged less than 18 years old. 2-Individuals with other autoimmune diseases (rheumatoid arthritis, dermatomyositis, connective tissue disease).

3-Congestive heart failure and presence of clubbing. 4-history of smoking. 5-Patients unable to co-operate for nail fold capillaroscopic examination.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cross sectional
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Nail fold capillary pattern changes in SSc patients | baseline